CLINICAL TRIAL: NCT03963141
Title: Retrospective Analysis to Describe Patient Profiles, Current Treatment Patterns and Economic Burden for Asthma Patients in UAE.
Brief Title: Retrospective Analysis to Describe Patient Profiles, Current Treatment Patterns and Economic Burden for Asthma Patients in UAE. A Descriptive Analysis of the Asthma Patient Population in the Emirate of Dubai With Respect to Healthcare Resource Utilization, Costs, and Asthma-related Treatment Pattern
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00139
Record Dates: First submitted 2019-04-03; First posted 2019-05-24 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Retrospective cohort study with an overall objective of to perform a descriptive analysis of the asthma patient population in the Emirate of Dubai with respect to healthcare resource utilization, costs, and asthma-related treatment patterns and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Minimum two claims with asthma diagnosis, 30 days apart, during the identification period
* Minimum 12 months of baseline period
* Age ≥ 18 years on the index date
* Continuous enrolment during the baseline period and at least 180 days of follow-up period; enrolment will be defined based on at least one activity during each 90-day period from the index date

Exclusion Criteria:

• Diagnosis of COPD during the baseline period. Diagnosis of COPD will be defined as ≥1 medical claim with an ICD-10 diagnosis in any position

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a diagnosis of asthma during the identification period will be considered for the analysis
Sampling Method: Non-Probability Sample
Enrollment: 40541 (Actual)
Dates: Start 2019-08-31 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Asthma Patients Number | 1 Year
  Number of unique asthma patients in the database during December 2015 through November 2018(summarized annually).it will be computed in the follow-up period and will be reported as a percentage and number of visits per person per year (PPPY). Utilization will be considered "all-cause" if the associated medical claim(s) has a diagnosis code in any position for any condition.
Asthma-related Cost | 1 Year
  Total asthma-related cost reported in the databse during December 2015 through November 2018(summarized annually).It will will be computed in the follow-up period and will be reported as a percentage and number of visits per person per year (PPPY). Utilization will be considered "asthma-related" if the associated medical claim(s) has ICD-10 diagnosis code for asthma as the principal diagnosis

SECONDARY OUTCOMES:
Asthma-related hopitalizations cost | 1 Year
  Number of asthma related hopistalizations and cost reported in the database during December 2015 through Novemebr 2018(Summairzed annually)
Astma-related prescription pattern | 1 Year
  Prescription pattern of asthma-related medication by drug class during December 2015 through November 2018
Severity of Asthma per total number of patients | 1 Year
  Number of patients classified as Mild, moderate and severe asthmatic patinets as per the international guidlines.

CONTACTS AND LOCATIONS:
Locations (1):
- Dha Claim, Dubai, United Arab Emirates

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00139&attachmentIdentifier=e13c29e1-6a21-4149-a9e2-54ec80673135&fileName=D2287R00139_Synopsis_Redacted_Clinical_Study_Report_(CSR)_RIMS_AZ_asthma.pdf&versionIdentifier=